CLINICAL TRIAL: NCT06376890
Title: Effects of Chili Pepper on Inflammation and Glycemic Control in Southern New Mexico
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New Mexico State University (Other)
Responsible Party: Principal Investigator, Peter Smoak, Assistant Professor, New Mexico State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Chile24
Record Dates: First submitted 2024-04-12; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Prediabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Intervention Model Description: A 3x2 model with 2 intervention groups (green and red chili) and a control group, and pre and post-intervention measures will be taken.
Who Masked: Participant
Masking Description: Only the primary investigator will know the intervention assigned to the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Red Chili Pepper (Experimental): 2.4 grams/day of red chili will be given to the red chili group for 10 weeks.
  Interventions: Dietary Supplement: Red chili peppers
- Green Chili Pepper (Experimental): 2.4 grams/day of green chili will be given to the green chili group for 10 weeks.
  Interventions: Dietary Supplement: Green Chili Pepper
- Placebo (Placebo Comparator): 2.4 grams/day of corn start will be given to the placebo group for 10 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Red chili peppers — 2.4 grams/day of powdered red chili pepper
  Arms: Red Chili Pepper
Dietary Supplement: Green Chili Pepper — 2.4 grams/day of powdered green chili peppers
  Arms: Green Chili Pepper
Dietary Supplement: Placebo — 2.4 grams of a metabolically equivalent placebo
  Arms: Placebo

SUMMARY:
Diabetes is a major health epidemic facing the United States and New Mexico. Currently, 11.6% of the US population (38.4 million) has diabetes, and 38.0% of US adults have prediabetes. It is estimated that around 70% of prediabetics will develop diabetes in their lifetime. In New Mexico, 48% of adults are at least prediabetic, and 12% of adults in southern New Mexico adults have diabetes. Moreover, major health disparities challenge the southern New Mexico region. Type 2 diabetes mellitus (T2DM) is generally linked with chronic inflammation, obesity, insulin resistance, and ultimately insulin dependence via pancreatic β-cell failure. Lessening pathological inflammation, a critically important factor that contributes to diabetes, can improve the disease. Furthermore, 89.8% of diabetics in the US are overweight or obese, this is a major risk for prediabetes and T2DM, as it causes insulin resistance and pancreatic β-cell dysfunction, Weight loss in people with T2DM and prediabetes has been demonstrated to affect glycemic control and metabolic parameters significantly. The purpose of this proposed study is to explore and establish the beneficial effects of 10 weeks of powdered chili pepper consumption on several parameters related to diabetes and prediabetes. This research will demonstrate how powdered chili pepper consumption can improve systemic inflammation, glycemic control, and body composition, and will provide valuable preliminary data for future funding to further examine these effects in Type 2 diabetics. This research is innovative because chili peppers are an already widely accepted food in Southern New Mexico. Demonstrating the beneficial improvements in diabetes-related markers using a popular food in the area may help to establish better treatments and protocols for an area that has health disparities. The first aim is to establish if 10 weeks of powdered red or green chili pepper consumption can significantly improve markers of inflammation, inflammatory capacity, and antioxidant capacity. The second aim is to establish if 10 weeks of powdered red or green chili pepper ingestion has a significant effect on resting blood glucose and insulin levels, connecting peptide (C-peptide) levels, and Homeostatic Model Assessment for Insulin Resistance (HOMA-IR). The third aim is to determine whether powdered chili pepper consumption for 10 weeks improves resting body composition and metabolic rate. This research is innovative because chili peppers are an already widely accepted food in Southern New Mexico. Demonstrating the beneficial improvements in diabetes-related markers using a popular food in the area may help to establish better treatments and protocols for an area with health disparities. Overall, this study will provide valuable insight and background knowledge for the use of chili peppers for the treatment of prediabetes and the prevention of diabetes progression.

ELIGIBILITY:
Inclusion Criteria:

* Must be eighteen years or older,
* Fasting blood glucose of 100mg/dl to 125mg/dl
* BMI of 24 or higher
* Must be willing to ingest powdered chili pepper
* Must be able to swallow tablets

Exclusion Criteria:

* Insulin dependent diabetes
* Thyroid disease
* History of metabolic disease
* Allergic to chili peppers
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Concentration of resting and fasted blood glucose measured in mg/dl | 10 Weeks
  Resting and fasted blood glucose will be measure at the pre- and post 10-week intervention time points. The outcome will be reported in mg/dl.
Concentration of resting and fasted insulin measured in pmol/L | 10 Weeks
  Resting and fasted blood glucose will be measure at the pre- and post 10-week intervention time points. The outcome will be reported in pmol/L
Concentration of circulating C-reactive protein reported as mg/dl. | 10 weeks
  Circulating concentrations of C-reactive protein (CRP) will be measured pre and post intervention and will be used as an indicator of whole-body inflammation. C-reactive protein will be reported in mg/dl.
Concentration of circulating interleukin (IL)-1 beta reported as pg/ml. | 10 weeks
  Circulating concentrations of IL-1 beta will be measured pre and post intervention and will be used as an indicator of inflammation and disease progression. IL-1 beta will be reported in pg/ml.
Concentration of circulating interleukin-6 (IL-6) reported as pg/ml. | 10 weeks
  Circulating concentrations of IL-6 will be measured pre and post intervention and will be used as an indicator of inflammation and disease progression. IL-6 will be reported in pg/ml.
Concentration of circulating interleukin tumor necrosis factor (TNF)-alpha reported as pg/ml. | 10 weeks
  Circulating concentrations of TNF-alpha will be measured pre and post intervention and will be used as an indicator of inflammation and disease progression. TNF-alpha will be reported in pg/ml.

SECONDARY OUTCOMES:
Concentration of circulating superoxide dismutase (SOD) reported as ng/ml. | 10 weeks
  Circulating concentrations super oxide dismutase will help to identify the effects of chili peppers on free radicals circulating in the body. SOD will be reported as ng/ml.
Concentration of circulating glutathione peroxidase reported as pg/ml. | 10 weeks
  Circulating concentrations glutathione peroxidase will help to identify the effects of chili peppers on free radicals circulating in the body. SOD will be reported as pg/ml.
Body composition measured as total fat mass and total fat free mass reported in kg. | 10 weeks
  Total fat mass and fat free mass will be measure in grams using the air displacement method. Body composition measured as total fat free and fat mass (kg) will help to understand if chili peppers have the ability to reduce total fat mass. Being overweight or obese is a contributor to metabolic diseases like diabetes and prediabetes.

IPD SHARING:
Plan to Share IPD: No
Individualized participant data will not be shared with anyone other than those on the research team.